CLINICAL TRIAL: NCT01163032
Title: A Multicenter, Randomized, Double-Mask, Placebo-Controlled, Parallel Study to Investigate the Efficacy and Safety of 20 mg Tasimelteon Versus Placebo in Totally Blind Subjects With N24HSWD Followed by an OLE Phase
Brief Title: Efficacy and Safety of Tasimelteon Compared With Placebo in Totally Blind Subjects With Non-24-Hour Sleep-Wake Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VEC-162-3201
Record Dates: First submitted 2010-07-02; First posted 2010-07-15 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Non-24-Hour Sleep-Wake Disorder
Keywords: Blindness; Eye Diseases; Nap Disorders; Circadian Rhythm Disorders; Sleep disorders; Circadian Rhythm Sleep Disorders; Dyssomnias; Nervous System Diseases
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Blindness; Eye Diseases; Chronobiology Disorders; Sleep Wake Disorders; Dyssomnias; Nervous System Diseases | interventions — tasimelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tasimelteon (Experimental): 20 mg tasimelteon capsules, PO daily for 6 months
  Interventions: Drug: tasimelteon
- placebo (Placebo Comparator): Placebo capsules, PO daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tasimelteon — 20 mg tasimelteon capsules, PO daily for 6 months
  Other Names: VEC-162
  Arms: tasimelteon
Drug: Placebo — Placebo capsules, PO daily for 6 months
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a six month double-mask treatment of tasimelteon or placebo in male and female subjects with Non-24-Hour Sleep-Wake Disorder

DETAILED DESCRIPTION:
Non-24-Hour Sleep-Wake Disorder (N24HSWD) occurs when individuals, primarily those without light perception, are unable to synchronize their endogenous circadian pacemaker to the 24-hour light-dark cycle, and the timing of their circadian rhythm instead reflects the intrinsic period of their endogenous circadian pacemaker. As a result, the circadian rhythm of sleep-wake propensity in these individuals moves gradually later and later each day if there circadian period is > 24 hours and earlier and earlier if < 24 hours. These individuals will be able to sleep well at night when their sleep-wake propensity rhythm is approximately aligned with the 24-hour light-dark and social cycle. However, after a short time, the endogenous sleep-wake propensity rhythm and the 24-hour light-dark cycle will move out of synchrony with each other, and they may have difficulty falling asleep until well into the night. In addition to problems sleeping at the desired time, the subjects experience daytime sleepiness and daytime napping.

This will be a multicenter, randomized, double-masked, placebo-controlled, parallel study. The study has two phases: the pre-randomization phase followed by either the randomization phase or the open-label extension (OLE). The pre-randomization phase comprises a screening visit where subject's initial eligibility will be evaluated, a circadian period (τ) estimation segment, and a variable-length in-phase transition segment in which subjects will wait to start treatment until their circadian phase is aligned with their target bedtime. Subjects that meet all entry criteria for the study will enter the randomization phase. During the randomization phase, subjects will be asked to take either 20 mg tasimelteon or placebo approximately 1 hour prior to their target bedtime for 26 weeks in a double-masked fashion. Subjects who have a τ greater than 24.0 and meet all entry criteria but that are ineligible for the randomization phase due to their τ estimate may be given the opportunity to participate in the OLE phase. During the OLE phase, subjects will take open-label 20mg tasimelteon for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability and acceptance to provide informed consent;
* No perception of light by the subject's own report;
* Diagnosis of N24HSWD as determined by:

  1. History (within the last 3 months) of trouble sleeping at night difficulty initiating sleep or staying asleep), difficulty awakening in the morning, or daytime sleepiness as determined by answering yes to at least one question in the Sleep Complaint Questionnaire and
  2. Urinary aMT6s demonstrates a progressive delay of the aMT6 acrophase time.
* Willing and able to comply with study requirements and restrictions including a commitment to a fixed 9-hour sleep opportunity during the study;
* Fluent in English;

Exclusion Criteria:

* Have a probable diagnosis of a current sleep disorder other than N24HSWD that is the primary cause of the sleep disturbance based on clinical investigator medical judgment;
* Current clinically significant cardiovascular, respiratory, neurologic, hepatic, hematopoietic, renal, gastrointestinal or metabolic dysfunction unless currently controlled and stable;
* History (within the 12 months prior to screening) of psychiatric disorders including Major Depressive Disorder, Generalized Anxiety Disorder, Axis II Disorders, delirium or any other psychiatric disorder that in the opinion of the clinical investigator would affect participation in the study or full compliance with study procedures;
* History of intolerance and/or hypersensitivity to melatonin or melatonin agonists;
* Worked night, rotating, or split (period of work, followed by break, and then return to work) shift work within 1 month of the screening visit or plan to work these shifts during the study;
* Unable to perform calls to the study IVR system to report questionnaire results;
* Exposure to any investigational drug, including placebo, within 30 days or 5 half lives (whichever was longer) of screening;
* Use of central nervous system prescription or OTC medications, other than melatonin, that affects the sleep-wake cycle
* Use of melatonin or melatonin agonist

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Vanda Pharmaceuticals
Locations (28):
- United States (23):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - SDS Clinical Trials Inc., Orange, California
  - VA Palo Alto Health Care System/PAIRE (San Fransisco Bay Area), Palo Alto, California
  - St. Johns Sleep Disorder Center - St. Johns Medical Plaza, Santa Monica, California
  - Radiant Research - Denver, Denver, Colorado
  - PAB Clinical Research Inc., Brandon, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Ocean Sleep Disorders Center - Ormond Beach, Ormond Beach, Florida
  - Sleep Disorders Center Of Georgia, Atlanta, Georgia
  - Suburban Lung Associates SC (Chicago Metropolitan Area), Elk Grove Village, Illinois
  - The Center for Sleep and Wake Disorders (Washington, D.C. Metropolitan Area), Chevy Chase, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Head-Pain Neurological Institute, Ann Arbor, Michigan
  - St. Luke's Sleep Medicine and Research Center (St. Louis Metropolitan Area), Chesterfield, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - Tri-State Sleep Disorders Center, Cincinnati, Ohio
  - Ohio Sleep Medicine Institute (Columbus Metropolitan Area), Dublin, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Columbia Research Group Inc., Portland, Oregon
  - Center For Sleep Medicine at Chestnut Hill Hospital, Philadelphia, Pennsylvania
  - Consolidated Clinical trials, Pittsburgh, Pennsylvania
  - SleepMed, Inc. - Columbia, Columbia, South Carolina
  - Todd J. Swick, M.D., P.A., Houston, Texas
- Germany (5):
  - Advanced Sleep Research GmbH, Berlin
  - Bergmannsheil University Hospital - Medical Clinic III, Bochum
  - Klinische-Forschung Hannover Mitte, Hanover
  - Universitaetsklinikum Glesen and Marburg gmbH/Schlaflabor - Sleep Lab University Marburg, Marburg
  - Bonomed Studiezentrum, Munich

REFERENCES:
- [Derived] Lockley SW, Dressman MA, Licamele L, Xiao C, Fisher DM, Flynn-Evans EE, Hull JT, Torres R, Lavedan C, Polymeropoulos MH. Tasimelteon for non-24-hour sleep-wake disorder in totally blind people (SET and RESET): two multicentre, randomised, double-masked, placebo-controlled phase 3 trials. Lancet. 2015 Oct 31;386(10005):1754-64. doi: 10.1016/S0140-6736(15)60031-9. Epub 2015 Aug 4. PMID 26466871

RESULTS

PARTICIPANT FLOW:
Recruitment Details: *Various category for the Randomization Phase: 4 patients in each treatment group discontinued due to study termination by the sponsor and 1 patient in the tasimelteon group discontinued due to travel across multiple time zones
Groups:
- Tasimelteon (Randomized); Open Label Tasimelteon: 20 mg tasimelteon capsules, PO daily for 6 months
  tasimelteon: 20 mg tasimelteon capsules, PO daily for 6 months
- Placebo (Randomized): Placebo capsules, PO daily for 6 months
  Placebo: Placebo capsules, PO daily for 6 months
Period: Randomization Phase
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized) | Open Label Tasimelteon
Started | 42 | 42 | 0 (Not applicable for Randomized Phase)
Completed | 32 | 30 | 0 (Not applicable for Randomized Phase)
Not Completed | 10 | 12 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0
Not completed — Adverse Event | 3 | 3 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Various* | 5 | 4 | 0
Not completed — Unsatisfactory Therapeutic Effect | 0 | 1 | 0
Period: Open Label Extension Phase
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized) | Open Label Tasimelteon
Started | 0 (Not applicable for Open Label Extension Phase) | 0 (Not applicable for Open Label Extension Phase) | 55 (3 randomized patients rolled into extension (2 randomized to tasimelteon and one to placebo))
Completed | 0 (Not applicable for Open Label Extension Phase) | 0 (Not applicable for Open Label Extension Phase) | 39
Not Completed | 0 | 0 | 16
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Study Termination | 0 | 0 | 7
Not completed — Unsatisfactory Therapeutic Effect | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 52 patients entered the OLE Phase from screening and 3 patients rolled over after completing the Randomization Phase (2:tasimelteon; 1:placebo). For this analysis, 3 patients are included in the randomized arms and not the OLE. A separate analysis has been done for both age and gender for the 3 subjects (Rand to OLE).
Groups:
- Total: Total of all reporting groups
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized) | Open Label Tasimelteon | Total
Number analyzed (Participants) | 42 | 42 | 52 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (12.63) | 50.7 (13.15) | 50.37 (13.17) | 50.6 (12.91)
Age, Customized [Mean (Standard Deviation); unit: years] — N = 2 (tasimelteon randomized then went to OLE) and 1 (placebo randomized then went to OLE)
  years
    Rand to OLE | 42.00 (5.66) | 54.00 (NA) — N = 1; Cannot be calculated | NA (NA) | 46.00 (8.00)
Sex/Gender, Customized [Number; unit: participants] — N = 2 (tasimelteon randomized then went to OLE) and 1 (placebo randomized then went to OLE)
  participants
    Rand to OLE (Female) | 0 | 0 | 0 | 0
    Rand to OLE (Male) | 2 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 25 | 60
  Male | 24 | 25 | 27 | 76

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Entrained as Assessed by Urinary aMT6
Description: Entrainment is a measure of synchronization of the master body clock to the 24-hour day. The circadian period (τ) was calculated using urinary aMT6s collected over four 48 hour periods , collected approximately 1 week apart for 4 separate weeks, during the screening and month 1 of the randomization phase of the trial. Entrainment was defined as having a post-baseline τ value less than 24.1 and a 95% CI that included 24.0.
Time Frame: 1 month
Population: Intent-to-Treat (ITT) Population: all subjects randomized into the study that have τ calculated post-randomization.
Measure: Number; unit: percentage of patients
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized)
Number analyzed (Participants) | 40 | 38
percentage of patients | 20 | 2.6

2. Primary Outcome: Proportion of Patients With a Clinical Response: Entrainment of aMT6 and Score of ≥ 3 on N24CRS
Description: Clinical response is defined as the coincident demonstration of entrainment (aMT6) and a score ≥ 3 on the Non-24 Clinical Response Scale (N24CRS). N24CRS measures improvement in sleep-wake measures and overall functioning (LQ-nTST, UQ-dTSD, MoST and CGI-C). Each assessment is scored as a 1 or 0 depending on the pre-specified threshold (see below).
  LQ-nTST: >45 minutes increase in average nighttime sleep duration; UQ-dTSD: >45 minutes decrease in average daytime sleep duration; MoST: >30 minutes increase and a standard deviation <2 hours during double-masked phase (6 months); CGI-C: <2.0 from the average of D112 and Day 183 compared to baseline
  For patients randomized to tasimelteon 20 mg and who also participated in the screening phase of Study 3203 (month 7 of treatment), the screening τ from Study 3203 was used if the patient did not become entrained in Study 3201 but did become entrained during the screening phase of Study 3203.
Time Frame: 6 months
Population: Analysis Population: all patients in the ITT population that had at least 70% of 1 circadian cycle of nighttime total sleep data reported during each phase (screening and post-randomization)
Measure: Number; unit: percentage of patients
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized)
Number analyzed (Participants) | 38 | 34
percentage of patients | 23.7 | 0

3. Other Pre Specified Outcome: Proportion of Patients With a Clinical Response: Entrainment of aMT6 and Score of ≥ 2 on N24CRS
Description: Clinical response is defined as the coincident demonstration of entrainment (aMT6) and a score ≥ 2 on the Non-24 Clinical Response Scale (N24CRS) which includes LQ-nTST, UQ-dTSD, MoST and CGI-C assessments. Each assessment is scored as a 1 or 0 depending on the pre-specified threshold (see below).
  LQ-nTST: >45 minutes increase in average nighttime sleep duration; UQ-dTSD: >45 minutes decrease in average daytime sleep duration; MoST: >30 minutes increase and a standard deviation <2 hours during double-masked phase (6 months); CGI-C: <2.0 from the average of D112 and Day 183 compared to baseline
  For patients randomized to tasimelteon 20 mg and who also participated in the screening phase of Study 3203 (month 7 of treatment), the screening τ from Study 3203 was used if the patient did not become entrained in Study 3201 but did become entrained during the screening phase of Study 3203.
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized)
Number analyzed (Participants) | 38 | 34
percentage of patients | 28.9 | 0

4. Other Pre Specified Outcome: Proportion of Patients With a Clinical Response (Score of ≥ 3 on N24CRS)
Description: Non-24 Clinical Response Scale (N24CRS) was a 4-item scale which includes LQ-nTST, UQ-dTSD, MoST and CGI-C assessments. Each assessment is scored as a 1 or 0 depending on the pre-specified threshold (see below).
  LQ-nTST: >45 minutes increase in average nighttime sleep duration; UQ-dTSD: >45 minutes decrease in average daytime sleep duration; MoST: >30 minutes increase and a standard deviation <2 hours during double-masked phase (6 months); CGI-C: <2.0 from the average of D112 and Day 183 compared to baseline
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized)
Number analyzed (Participants) | 38 | 34
percentage of patients | 28.9 | 2.9

5. Secondary Outcome: Proportion of Patients Entrained as Assessed by Urinary Cortisol
Description: Entrainment is a measure of synchronization of the master body clock to the 24-hour day. The circadian period (τ) was calculated using urinary cortisol collected over four 48 hour periods, approximately 1 week apart for 4 separate weeks, during the screening and month 1 of the randomization phase of the trial. Entrainment was defined as having a post-baseline τ value less than 24.1 and a 95% CI that included 24.0.
Time Frame: 1 month
Population: Intent-to-Treat (ITT) Population: all subjects randomized into the study that have τ calculated post-randomization.
Measure: Number; unit: percentage of patients
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized)
Number analyzed (Participants) | 40 | 38
percentage of patients | 17.5 | 2.6

6. Secondary Outcome: Average Clinical Global Impression of Change (CGI-C)
Description: CGI-C scores range from 1 (very much improved) to 7 (very much worse). The average post-randomization score was obtained for each patient by averaging the last 2 scheduled assessments (Day D112 and Day D183). Lower number indicates improvement.
Time Frame: Day 112 and 183
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized)
Number analyzed (Participants) | 38 | 34
score | 2.6 (0.20) | 3.4 (0.21)

7. Secondary Outcome: Proportion of Responders With a Combined Sleep/Wake Response for LQ-nTST (≥ 90 Minutes) and UQ-dTSD (≤ 90 Minutes)
Description: The sleep/wake response represents measurement of the combined improvement in the nighttime sleep duration and daytime sleep duration. Individuals that have an improvement in nighttime sleep and daytime sleep, defined as an increase of 90 minutes or more in the lower quartile of subjective nighttime total sleep time (LQ-nTST) and a decrease of 90 minutes or more in the upper quartile of daytime total sleep duration (UQ-dTSD) are considered to be a responder.
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized)
Number analyzed (Participants) | 38 | 34
percentage of patients | 13.2 | 2.9

8. Secondary Outcome: Average Lower Quartile of Nights of Nighttime Total Sleep Time (LQ-nTST)
Description: LQ-nTST measures the difference in average nighttime sleep during the patient's worst 25% of nights (shortest total nighttime sleep) between the randomized phase (6 months)and the screening phase (~ 6 weeks). The higher number indicates improvement.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized)
Number analyzed (Participants) | 38 | 34
minutes | 56.80 (9.305) | 17.08 (9.702)

9. Secondary Outcome: Average Upper Quartile of Days of Subjective Daytime Sleep Duration (UQ-dTSD)
Description: UQ-dTSD measures the difference in average daytime sleep during the patient's worst 25% of days (longest total daytime sleep) between the randomized phase (6 months) and the screening phase (~ 6 weeks). Lower number indicates improvement.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized)
Number analyzed (Participants) | 38 | 34
minutes | -46.48 (6.595) | -17.87 (6.889)

10. Secondary Outcome: Average Midpoint of Sleep (MoST)
Description: Midpoint of Sleep Timing (MoST) is the measurement of the average midpoint of sleep time relative to bedtime. The average MoST value will trend to 0 as an individual's sleep becomes more fragmented. Improvement is defined as an increase in the average.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized)
Number analyzed (Participants) | 38 | 34
minutes | 35.00 (5.313) | 14.48 (5.547)

11. Post Hoc Outcome: Proportion of Responders With a Combined Sleep/Wake Response for LQ-nTST (≥ 45 Minutes) and UQ-dTSD (≤ 45 Minutes)
Description: Responder analysis with responder defined as an increase of 45 minutes or more in (LQ-nTST) and a decrease of 45 minutes or more in (UQ-dTSD).
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized)
Number analyzed (Participants) | 38 | 34
percentage of patients | 31.6 | 8.8

12. Other Pre Specified Outcome: Proportion of Patients With a Clinical Response (Score of ≥ 2 on N24CRS)
Description: as for outcome 4
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized)
Number analyzed (Participants) | 38 | 34
percentage of patients | 57.9 | 20.6

13. Secondary Outcome: Number of Patients With a Treatment Emergent Adverse Event (Open Label Extension Phase Only)
Description: Adverse events were recorded in the source documents from the time of the patient's informed consent signature until the end of the patient's study participation. An AE was defined as any untoward medical occurrence in a clinical investigation patient who does not necessarily have causal relationship with treatment.
Time Frame: 6 months
Population: One subject who rolled into the OLE from the randomized phase (tasimelteon) experienced an unrelated TEAE during the OLE phase.
Measure: Number; unit: participants
Arm/Group | Open Label Tasimelteon
Number analyzed (Participants) | 54
participants | 37

ADVERSE EVENTS:
Time Frame: 1st dose to 30 days following last administration of study treatment
Description: 55 subjects enrolled into the Open Label phase (including 3 randomized subjects who rolled into the OLE). One subject enrolled in the Open Label phase but did not take any study drug.
Arm/Group | Tasimelteon (Randomized) | Placebo (Randomized) | Open Label Tasimelteon
Serious Adverse Events (participants affected / at risk) | 4/42 | 2/42 | 2/54
Other Adverse Events (participants affected / at risk) | 20/42 | 13/42 | 21/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasimelteon (Randomized) (N=42) | Placebo (Randomized) (N=42) | Open Label Tasimelteon (N=54)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Serotonin Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasimelteon (Randomized) (N=42) | Placebo (Randomized) (N=42) | Open Label Tasimelteon (N=54)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 5 (6)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 5 (6)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (2) | 2 (2)
Asparate aminotransferase increased (Investigations) | 3 (3) | 2 (2) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 7 (11) | 3 (3) | 4 (4)
Abnormal dreams (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 3 (3) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No